CLINICAL TRIAL: NCT02598063
Title: A Randomized, Open-label Study Evaluating the Efficacy and Safety of Peginterferon Alfa-2a (40KD) (PEGASYS®) or Adefovir Dipivoxil (ADV) in Patients With Lamivudine-resistant HBeAg Positive Chronic Hepatitis B
Brief Title: A Study to Evaluate Efficacy and Safety of Peginterferon Alfa-2a (Pegasys) and Adeforvir Dipivoxil (ADV) in Participants With Lamivudine-Resistant Hepatitis B e Antigen (HBeAg)-Positive Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18376
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; Lamivudine; peginterferon alfa-2a

ARMS (2):
- ADV + Lamivudine (Active Comparator): Participants will receive ADV and lamivudine tablets at a dose of 10 mg orally QD for first 12 weeks followed by ADV for 60 weeks.
  Interventions: Drug: Adefovir dipivoxil; Drug: Lamivudine
- Peginterferon alfa-2a + Lamivudine (Experimental): Participants will receive peginterferon alfa-2a injection at a dose of 180 micrograms (mcg) once weekly (QW) and 100 milligrams (mg) lamivudine tablets orally once daily (QD) for first 12 weeks followed by peginterferon alfa-2a for 36 weeks.
  Interventions: Drug: Lamivudine; Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Adefovir dipivoxil — ADV will be administered orally at a dose of 10 mg QD for 72 weeks.
  Arms: ADV + Lamivudine
Drug: Lamivudine — Lamivudine tablets will be administered orally at a dose of 10 mg QD for 12 weeks.
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a injection will be administered at a dose of 180 mcg QW for 48 weeks.
  Other Names: Pegasys
  Arms: Peginterferon alfa-2a + Lamivudine

SUMMARY:
This study will evaluate the efficacy and safety of peginterferon alfa-2a or ADV, in participants with lamivudine-resistant HBeAg-positive chronic hepatitis B. Participants will be randomized to receive either peginterferon alfa-2a for 48 weeks in combination with oral lamivudine for the first 12 weeks, or ADV for 72 weeks in combination with oral lamivudine for the first 12 weeks. The anticipated time on study treatment is 72 weeks, and the target sample size is 255 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants 18-65 years of age
* Hepatitis B surface antigen (HBsAg)-positive, HBeAg-positive, and anti-HBs-negative for greater than or equal to (>=) 6 months
* Receiving lamivudine currently, and for >=6 months
* hepatitis B virus (HBV)-deoxyribonucleic acid (DNA) decreased >=2 log during lamivudine treatment on >=1 occasion
* Absence of cirrhosis confirmed by liver biopsy in previous 6 months

Exclusion Criteria:

* Other drugs with activity against HBV within the prior 6 months, except lamivudine
* Antiviral, anti-neoplastic, or immunomodulatory therapy less than or equal to (<=) 6 months before study - Active infection with hepatitis A, C, or D virus, or human immunodeficiency virus
* Decompensated liver disease
* Medical condition associated with another chronic liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2005-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
HBeAg seroconversion (defined as loss of HBeAg and presence of anti-HBe) at Week 72 | Week 72

SECONDARY OUTCOMES:
Loss of HBeAg | Week 48, and 72
Reduction in hepatitis B virus deoxyribonucleic acid (HBV DNA) | Week 48, and 72
Alanine transaminase (ALT) normalization | Week 48, and 72
Hepatitis B surface antigen (HBsAg) seroconversion | Week 48, and 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (7):
- China (6):
  - Beijing
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Jinan
  - Shanghai
- Hong Kong, Hong Kong